CLINICAL TRIAL: NCT05079971
Title: The EAGLET Project: EEG vs aEEG to Improve the Diagnosis of neonataL Seizures and Epilepsy - a Randomised Trial
Brief Title: EAGLET: EEG vs aEEG to Improve the Diagnosis of neonataL Seizures and Epilepsy
Acronym: EAGLET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Luton and Dunstable Hospital NHS Foundation Trust (Unknown); Infant, University College Cork, Ireland (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ronit Pressler, Dr (Clinical Neurophysiology), Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: A 096043
Record Dates: First submitted 2021-09-13; First posted 2021-10-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Seizures
Keywords: Neonatal Seizures; cEEG; aEEG; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A is a control group with aEEG monitoring only, and with retrospective cEEG review (Active Comparator)
  Interventions: Diagnostic Test: Group B: aEEG with concurrent multichannel (full) continuous cEEG review by clinical neurophysiology
- Group B is undergoing aEEG monitoring with concurrent full EEG review (Experimental)
  Interventions: Diagnostic Test: Group B: aEEG with concurrent multichannel (full) continuous cEEG review by clinical neurophysiology

INTERVENTIONS:
Diagnostic Test: Group B: aEEG with concurrent multichannel (full) continuous cEEG review by clinical neurophysiology — In group B, the standart-care equivalent aEEG review is undertaken by NICU staff via a 2-channel display. In addition to the standard care, concurrent full EEG is reviewed remotely with regular feedback by a specialist trained clinical neurophysiologist. The clinical neurophysiology reports only on seizure burden, no information or direction is provided regarding clinical management.

SUMMARY:
The current project undertakes a prospective multicentre randomised controlled trial to evaluate whether full or continuous electroencephalography (cEEG) is superior to amplitude-integrated electroencephalography (aEEG) in the real time evaluation and diagnosis of neonatal seizures and in reducing time to treatment. At-risk new-born infants will be recruited on the participating neonatal intensive care units (NICUs) by trained specialist staff and will have 24 hours of EEG monitoring.

DETAILED DESCRIPTION:
Seizures are the most common neurological emergency in the neonatal period, affecting over 2000 infants per year in the UK. Although neonatal seizures usually result from acute brain insults, about 10-15% represent genetic forms of epilepsy which are often diagnosed late, thus limiting the timely use of targeted therapies. Lack or delayed initiation of treatment results in a high seizure burden which is independently associated with worse clinical outcomes.

Diagnosing neonatal seizures is challenging because most have only subtle or no clinical manifestation. The gold standard for seizure detection is continuous electroencephalography (cEEG). cEEG can assist with establish the aetiology of seizures, and their management. However, this capability is lacking in most neonatal intensive care units (NICU) due to lack of on-site specialist support. The more common amplitude-integrated EEG (aEEG) uses a limited number of electrodes and is easier to apply and interpret but has been shown to miss a significant number of seizures. It is unclear how often seizure treatment is missed or delayed due to lack of cEEG access. Although studies have compared the diagnostic value of aEEG and cEEG retrospectively, the measured sensitivity of aEEG ranges widely (25-85%), likely due to poor design (retrospective, lack of adequate control group, no power calculations).

The current project undertakes a prospective multicentre randomised controlled trial to evaluate whether cEEG is superior to aEEG in the real time evaluation and diagnosis of neonatal seizures and in reducing time to treatment. At-risk neonates will be recruited on the NICU by trained specialist staff and will have 24 hours of EEG monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Term or preterm neonate, born at post-menstrual age (PMA) 32-44 weeks;
2. And at least one of the following:

   (2.1) Neonate with any clinical event suspicious of seizures (2.2) Neonate at high-risk of seizures with confirmed or suspected: (2.2.1) Hypoxic ischaemic encephalopathy (moderate to severe, or deemed eligible for therapeutic hypothermia) (2.2.2) Cerebral vascular insult (e.g., perinatal arterial ischaemic stroke, cerebral venous sinus thrombus) (2.2.3) Meningitis / encephalitis - Inflammatory (2.2.4) Inborn error of metabolism (2.2.5) Brain malformation (2.2.6) Large intraventricular haemorrhage (III-IV)
3. Infant is up to 28 days of age
4. Written informed parental consent can be obtained.

Exclusion Criteria:

1. No parental consent
2. Poor prognosis of immediate survival
3. Any contraindication to perform EEG (e.g. structural pathologies interfering with EEG electrode placement, such as cephalohematoma or subgaleal haemorrhage).
4. Infants born at less than 31+6 weeks PMA and infants who are or are suspected to be experiencing or are at high-risk of seizures when aged 29 days or older.

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Seizure detection yield of aEEG compared to full EEG | Each participant will be assessed in Group A (aEEG review only) or Group B (a+cEEG) for 24 hours.
  The primary outcome measure for the study is the difference in the number of correctly identified seizures by NICU staff in real time with (full EEG) or without (aEEG only) the support of clinical neurophysiology.

SECONDARY OUTCOMES:
Time from first recorded seizure to first recognised seizure and to treatment. | Each participant's seizure burden, treatment and discharge timelines will be recorded up until their discharge from the hospital, or for up to 6 months, whichever came first.
  Their time to treatment and time to discharge will also be noted.
Number of false positive seizure detections clinically and/or by aEEG | Followed until their discharge from hospital, or for up to 6 months, whichever came first.
Off-line seizure burden (min/hr) detected by aEEG vs detected by cEEG | Followed until their discharge from hospital, or for up to 6 months, whichever came first.
Parental and staff acceptance of EEG monitoring (combined cohort) using questionnaire. | Parents may fill in the questionnaire online after their infant's discharge from hospital, the questionnaire will take a maximum of 10 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pinchefsky EF, Hahn CD. Outcomes following electrographic seizures and electrographic status epilepticus in the pediatric and neonatal ICUs. Curr Opin Neurol. 2017 Apr;30(2):156-164. doi: 10.1097/WCO.0000000000000425. PMID 28118303
- [Background] Malone A, Ryan CA, Fitzgerald A, Burgoyne L, Connolly S, Boylan GB. Interobserver agreement in neonatal seizure identification. Epilepsia. 2009 Sep;50(9):2097-101. doi: 10.1111/j.1528-1167.2009.02132.x. Epub 2009 Jun 1. PMID 19490044
- [Background] Boylan GB, Kharoshankaya L, Mathieson SR. Diagnosis of seizures and encephalopathy using conventional EEG and amplitude integrated EEG. Handb Clin Neurol. 2019;162:363-400. doi: 10.1016/B978-0-444-64029-1.00018-7. PMID 31324321
- [Background] Pellegrin S, Munoz FM, Padula M, Heath PT, Meller L, Top K, Wilmshurst J, Wiznitzer M, Das MK, Hahn CD, Kucuku M, Oleske J, Vinayan KP, Yozawitz E, Aneja S, Bhat N, Boylan G, Sesay S, Shrestha A, Soul JS, Tagbo B, Joshi J, Soe A, Maltezou HC, Gidudu J, Kochhar S, Pressler RM; Brighton Collaboration Neonatal Seizures Working Group. Neonatal seizures: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2019 Dec 10;37(52):7596-7609. doi: 10.1016/j.vaccine.2019.05.031. No abstract available. PMID 31783981
- [Background] Gossling L, Alix JJP, Stavroulakis T, Hart AR. Investigating and managing neonatal seizures in the UK: an explanatory sequential mixed methods approach. BMC Pediatr. 2020 Jan 28;20(1):36. doi: 10.1186/s12887-020-1918-4. PMID 31992265
- [Background] Rakshasbhuvankar A, Paul S, Nagarajan L, Ghosh S, Rao S. Amplitude-integrated EEG for detection of neonatal seizures: a systematic review. Seizure. 2015 Dec;33:90-8. doi: 10.1016/j.seizure.2015.09.014. Epub 2015 Sep 26. PMID 26456517